CLINICAL TRIAL: NCT01965613
Title: A Phase II Open Label Study of Xilonix in Subjects With Pyoderma Gangrenosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-PT025
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pyoderma Gangrenosum
Keywords: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — bermekimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label-Xilonix (Experimental): Open label-Xilonix
  Interventions: Biological: Xilonix

INTERVENTIONS:
Biological: Xilonix — IV

SUMMARY:
The purpose of this study is to determine if treatment with Xionix will improve wound healing for patients with pyoderma gangrenosum.

DETAILED DESCRIPTION:
XBiotech owned bermekimab and sponsored and completed study prior to Dec 30, 2019.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18
2. History of pyoderma gangrenosum with or without other systemic disease.

Exclusion Criteria:

1. Treatment with any biologicals (including intravenous immunoglobulin) or investigational agents within the last 4 weeks (or 5 half-lives, whichever is longer).
2. Treatment with corticosteroids or cyclosporine within the last 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Physician's Wound Assessment & Patient's Global Assessment | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- XBiotech Investigative Site, Tallahassee, Florida, United States